CLINICAL TRIAL: NCT05794672
Title: A Phase 1, Randomised, Single-blind, Placebo-controlled, Single-centre Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of Elarekibep Given Twice Daily as Inhaled or a Single IV Formulation in Healthy Japanese Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Elarekibep in Healthy Japanese Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This decision was based on lung findings from a non-clinical 13-week GLP toxicology study, which are not a concern for the active clinical studies but do not support long-term use and progression to later-stage development.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2912C00002; 2022-000426-22 (EudraCT Number)
Record Dates: First submitted 2023-02-20; First posted 2023-04-03 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Healthy Subjects (Indication: Asthma)
Keywords: Heterogenous respiratory disease; Pulmonary inflammation; Healthy subjects; Japanese subjects; Interleukin 4 receptor alpha antagonist
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Part A1: Each subject in three of the single inhaled dose cohorts will receive a single inhaled dose A, B, or C elarekibep and placebo in the fourth cohort.
  Part A2: Each subject will receive a single Intravenous (IV) dose D elarekibep in one cohort.
  Interventions: Drug: Elarekibep; Drug: Placebo
- Part B (Experimental): Each subject will receive multiple inhaled doses C elarekibep or placebo twice daily (BID) for 6 days in the first cohort and a single inhaled dose on Day 7 in the second cohort.
  Interventions: Drug: Elarekibep; Drug: Placebo

INTERVENTIONS:
Drug: Elarekibep — Subjects will receive single or multiple inhaled doses A, B or C, or single IV dose D of elarekibep.
  Other Names: AZD1402
Drug: Placebo — Subjects will receive single or multiple inhaled doses A, B or C.

SUMMARY:
This study will assess the safety, tolerability and pharmacokinetics (PK) of elarekibep after single and multiple doses given twice daily (BID) by inhalation or intravenous (IV) in healthy Japanese subjects compared with placebo.

DETAILED DESCRIPTION:
This is a Phase I, randomised, single-blind, placebo-controlled, single-centre study. This study comprises upto a total of 42 subjects.

This study consists of two parts: A single dose part (Part A1 and Part A2) and a multiple dose part (Part B).

Part A and Part B will comprise of the following:

* Each subject will be involved in the study for up to 9 weeks if enrolled in Part A and up to 10 weeks if enrolled in Part B.
* A screening period of maximum 28 days.
* Treatment period: Part A: Study treatment Day 1; Part B: Study treatment Days 1 to 6 and a single inhaled dose on Day 7.
* A safety follow-up call will be conducted 7 (± 1) days after elarekibep or placebo administration.
* A safety follow-up visit will be conducted 30 (± 2) days after elarekibep or placebo administration in each cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be aged 20 to 55 years.
* Subject must have a Body Mass Index (BMI) between 18 and 35 kg/m2 and weigh a minimum of 48 kg.
* First generation subjects who were born in Japan and who have both parents and grandparents of Japanese descent.
* All females must have a negative pregnancy test at the Screening Visit (serum) and on admission (urine) to the Clinical Unit and must not be lactating or planning to become pregnant.
* Subjects who are non-smokers or ex-smokers who have smoked no more than twice in the 3 months preceding the first dose of study drug.
* Must be able to demonstrate proper inhalation technique using the monodose Dry Powder Inhaler (DPI) device.
* Able to perform acceptable pulmonary function testing for Forced Expiratory Volume in one second (FEV1) according to American Thoracic Society (ATS)/European Respiratory Society (ERS) acceptability criteria.

Exclusion Criteria:

* History or clinical manifestations of any clinically significant medical disorder which may either put the subject at risk because of participation in the study, influence the results, or affect the subject's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease.
* Any clinically significant illness, infection, medical/surgical procedure, or trauma within 4 weeks of Day 1 or planned in-patient surgery or hospitalization during the study period.
* Diagnosis of Sjögren's syndrome.
* Any laboratory values with deviations from the study's laboratory parameters.
* Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and Human Immunodeficiency Virus (HIV).
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting Electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG.
* Known or suspected history of drug abuse in the last 5 years.
* Known or suspected history of alcohol abuse or excessive intake of alcohol in the last 2 years.
* Positive screen for drugs of abuse, alcohol or cotinine at the Screening Visit.
* History of anaphylaxis following any biologic therapy or vaccine and known history of allergy or reaction to any component of the Investigational Medicinal Product (IMP) formulation.
* Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 450 mL during the 3 months prior to the Screening Visit.
* Excessive intake of caffeine containing drinks or food.
* Participation in more than 4 clinical studies with IMPs in the last year.
* Involvement of subjects who have a significant history of recurrent or ongoing dry eye syndrome of any cause that may be chronic or acute and that may affect the interpretation of safety data associated with the potential for ADAs targeted to elarekibep.
* Subjects with a positive diagnostic nucleic acid test (using Polymerase Chain Reaction [PCR]) and/or rapid antigen test for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) at screening and up to randomisation.
* Diagnosis of/suspected COVID-19 infection with associated pneumonia/pneumonitis.
* Receipt of COVID-19 vaccine (vaccine or booster dose) within 30 days prior to randomisation.
* History of anaphylaxis to any biologic therapy or vaccine.
* History of hypersensitivity that required the use of epinephrine or hospitalization.
* Known history of allergy or reaction to any component of the IMP formulation.
* History of allergic conjunctivitis and/or dry eye syndrome.
* Clinically significant lower respiratory tract infection not resolved within 4 weeks prior to screening.
* History of cancer within the last 10 years except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix treated and considered cured. Any history of lymphoma is not allowed.
* Males who are sexually active with a female partner of childbearing potential and who have not had a vasectomy and who do not agree to comply with highly effective methods of contraception from Day 1 until 90 days after the last dose of IMP.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2023-07-08 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events | Up to Follow-up [Part A: 60 days, Part B: 67 days)
  The safety and tolerability of elarekibep after single and multiple inhaled or single Intravenous (IV) dose administrations in healthy Japanese subjects will be assessed.
Collection of blood samples for the measurement of safety immunobiomarkers | Part A: Screening (Day -28) to Day 3; Part B: Screening (Day -28 to -2) to Follow-up ([Day 37 ± 2)]
  The safety and tolerability of elarekibep after single and multiple inhaled or single Intravenous (IV) dose administrations in healthy Japanese subjects will be assessed.

SECONDARY OUTCOMES:
Maximum observed serum (peak) drug concentration [Cmax] | Part A: Day 1 to Day 3, Part B: Day 1 to Day 9
  The Cmax of elarekibep after single and multiple inhaled or single IV doses in healthy Japanese subjects will be evaluated.
Area under the serum concentration curve from zero to the last quantifiable concentration (AUClast) | Part A: Day 1 to Day 3, Part B: Day 1 to Day 9
  The AUClast of elarekibep after single and multiple inhaled or single IV doses in healthy Japanese subjects will be evaluated.
Area under serum concentration time curve from zero to infinity (AUCinf) | Day 1
  The AUCinf of elarekibep after single and multiple inhaled or single IV doses in healthy Japanese subjects will be evaluated.
Presence of elarekibep Antidrug Antibody (ADA) | Part A: Day 1; Part B: Day 1, Day 14 to Follow-up/ETV ([Day 37 ± 2)
  The immunogenicity of elarekibep in healthy Japanese subjects will be evaluated.
Standardised taste questionnaires | Part A: Day 1, Part B: Day 1
  Taste characteristics will be assessed within 5 minutes from dosing. There are 10 questions each of which is scored on a scale of 0 to 10 where 0 is the low range while 10 is the extreme range.
  Palatability will be assessed as measured by taste scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home